CLINICAL TRIAL: NCT00471029
Title: Compare Gastric Acid Suppression of Esomeprazole by Oral or Intravenous Administration - A Randomized Trial
Brief Title: Compare Efficacy of Gastric Acid Suppression by Oral and Intravenous Administration of Esomeprazole in Patients With Peptic Ulcer
Acronym: NPH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pamela Youde Nethersole Eastern Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKEC-2005-110
Record Dates: First submitted 2007-05-08; First posted 2007-05-09 (Estimated); Last update posted 2007-05-09 (Estimated); Status verified 2007-05

CONDITIONS: Peptic Ulcer
Keywords: pH study, peptic ulcer, proton pump inhibitor
MeSH Terms: conditions — Peptic Ulcer | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: esomeprazole

SUMMARY:
The purpose of this study is to compare the gastric acid suppression profile among different regimen (Oral Vs Intravenous)of administration of proton pump inhibitor - Esomeprazole by 24hours intragastric pH monitoring.

DETAILED DESCRIPTION:
Peptic ulcer bleeding is a common medical emergency. Although primary hemostasis can be achieved by endoscopic hemostasis in more than 90% of cases, rebleeding during the first 72 hours is still common. The use of secretory inhibitors in ulcer bleeding had theoretical benefit in preventing rebleeding. In vitro, platelet aggregation and disaggregation, coagulation and fibrinolysis are strongly dependent on intra-gastric pH. When pH falls below 6.0, platelet disaggregation takes place and below 4.0, fibrin clots dissolved. Pharmacological studies have clearly shown that primed proton-pump inhibitor (PPI) infusion is superior to H2-receptor blocler (H2B) injection or infusion in maintaining high intra-gastric pH. Randomized trials had demonstrated the advantage of adjuvant use of intravenous or oral PPI in reducing rebleeding as compared to placebo. However, as Asian subjects generally have lower body weight and acid output than Caucasians, the dosage of PPI required for prevent rebleeding may be different. Lin et al had demonstrated that in an Asian population study, in order to show a significant clinical effect in prevent peptic ulcer rebleeding after endoscopic hemostasis, at least a 30% difference in duration in maintaining an intragastric pH >6 must be achieved. As there is substantial cost implication of routine use of high dose intravenous PPI infusion (80mg bolus + 8mg/hour for 72 hours, cost ~HKD$1100) against high dose oral esomeprazole (40mg BD for 3 days, cost ~HKD$60), the optimal doses and routes of administration of PPI in achieving effective acid suppression is needed to be clearly defined.

Protocol:

Patients presented with bleeding peptic ulcers (melena, hememtesis) will undergo endoscopy. If clean base peptic ulcer which dos not require endoscopic treatment is diagnosed, consented patients will randomly allocated into 2 groups using sealed envelopes containing a therapeutic option derived from a randomized table.

1. Esomeprazole infusion (80mg bolus then 8mg/hour) (192mg/d)
2. Esomeprazole Tablet oral 40mg 12 hourly (80mg/d)

A pH electrode with internal reference (Synetic) was inserted transnasally and positioned 10cm below the cardia. It was calibrated before and after the pH recording with standard buffer solutions of pH 7.00 and pH 1.00. The electrode was connected to a data logger (Mircodigitrapper, Synetic). At the end of 24hours recording, the data were transfer to a personal computer for analysis. Medication will be given after insertion of intra-gastric pH monitor probe.

Outcome measures Primary Outcome: total % Time pH > 6 & 4 Secondary outcome: Median intragastric pH & Time to reach pH 4 and 6

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-bleeding peptic ulcer which do not require endoscopic therapy.
2. Chinese, Age ³18 and <90
3. Provision of an informed written consent signed by the patient.

Exclusion Criteria:

1. Treatment of antisecretory drugs during the preceding 4 weeks
2. The present inter-current ulcer complication (gastric outlet obstruction or ulcer perforation)
3. Presence of esophageal / gastric varices
4. aspirin or NSAID user
5. Pregnancy
6. Age <18 or >90
7. Moribund patients, patients with severe liver or renal disease
8. Known sensitivity to proton pump inhibitors
9. Previous gastric surgery (except simple patch repair)
10. Patient unable to give written consent
11. Special population, e.g. prisoner, mentally disabled, investigators' student or employees

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-09; Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
percentage of time intragstric pH > 6 and > 4 | 24hours after endoscopy

SECONDARY OUTCOMES:
Median intragastric pH | 24hours after endoscopy
time to attain intragastric pH 4 & 6 | 24hours after endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Simon K.H. Wong, MBChB, FRCSEd, FHKAM, Principal Investigator — Pamela Youde Nethersole Hospital - Surgery; Michael K.W. Li, MD, Study Chair — PYNEH
Locations (1):
- Pamela Youde Nethersole Eastern Hospital, Hong Kong, China